CLINICAL TRIAL: NCT06557720
Title: Exploring the Characteristics of Epileptogenic Foci in Drug-Resistant Epilepsy Using Multimodal Imaging Techniques: A Prospective Observational Cohort Study
Brief Title: Exploring the Characteristics of Epileptogenic Foci in Drug-Resistant Epilepsy Based on Multimodal Imaging Technology
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20242168
Record Dates: First submitted 2024-08-01; First posted 2024-08-16 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-06

CONDITIONS: Drug Resistant Epilepsy; Magnetic Resonance Imaging; Electroencephalogram (EEG)
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intractable epilepsy patients.: Based on the hybrid fusion technology of PET-fMRI-EEG, this study explores the characteristics of brain network damage in refractory epilepsy, identifies key network nodes (such as central nodes), and provides more assistance for the diagnosis of drug-resistant epilepsy.

SUMMARY:
Using multimodal imaging technology, this study aims to explore the characteristics of epileptogenic foci in patients with drug-resistant epilepsy and identify key network nodes (such as central nodes) to provide more assistance for the diagnosis of drug-resistant epilepsy.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study. It prospectively recruited 50 patients with drug-resistant epilepsy from the Epilepsy Center of the Department of Neurology at Xijing Hospital, all aged 18 years or older. It collected general information and clinical baseline data such as magnetic resonance imaging; gathered multimodal imaging data once; analyzed the characteristics of epileptogenic foci in patients with drug-resistant epilepsy; and performed statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old;
2. Meet the 2010 International League Against Epilepsy (ILAE) diagnostic criteria for drug-resistant epilepsy;
3. Duration of epilepsy ≥2 years, with an average seizure frequency of ≥2 times per month in the 3 months prior to enrollment;
4. Adequate intake of two or more anti-epileptic drugs, with no intervention in the treatment plan during the trial period;
5. Capable of cooperating to complete treatment and related examination items; The patient and family fully understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. In a state of continuous epileptic seizures;
2. Complicated with severe infections, cerebrovascular diseases, malignant tumors, and other diseases, accompanied by severe dysfunction of the heart, liver, kidney, or other organs, or with mental disorders, or with uncorrectable hyperglycemia, or 3.patients on long-term use of corticosteroid medications;

4.Pregnant or lactating women; 5.Contraindications for PET, MR, EEG examinations; 6.Patients with examinations (with ferromagnetic metal implants in the body; high fever); 7.Participating in other clinical trials at the same time; 8.The patient or family withdraws the informed consent form.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: drug-resistant epilepsy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2027-06-11 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The characteristics of hybrid imaging in patients with different types of refractory epilepsy. | baseline
  Based on PET-FMRI-EEG hybrid fusion technology, explore the brain network characteristics of epilepsy patients.PET detects areas of reduced glucose metabolism, using radioactive isotopes (such as 18F-labeled fluorodeoxyglucose) to reflect the glucose metabolism of brain tissue. Typically in epilepsy patients, areas of hypometabolism may indicate the presence of epileptic foci. By using fMRI or EEG data, the synchronization of activities between different brain regions is analyzed to understand the organization and functional connectivity patterns of the brain network.
The characteristics of PET, fMRI, and EEG indicators in patients with different types of intractable epilepsy. | baseline
  Using different data analysis methods to explore the characteristics of PET, fMRI, and EEG indicators in patients with various types of intractable epilepsy.The characteristics of the power spectrum of various EEG frequency bands (Delta, Theta, Alpha, Beta, Gamma waves) and brain functional connectivity.

SECONDARY OUTCOMES:
Quality of Life in Epilepsy 31 (QOLIE-31) | baseline，4weeks
  It assesses various aspects of a patient's life that can be affected by their condition, including physical, emotional, and social well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wen, Study Chair — Xi Jing hospital
Locations (1):
- Xijing Hospital of Air Force Military Medical University, Xi'an, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forsgren L, Beghi E, Oun A, Sillanpaa M. The epidemiology of epilepsy in Europe - a systematic review. Eur J Neurol. 2005 Apr;12(4):245-53. doi: 10.1111/j.1468-1331.2004.00992.x. PMID 15804240
- [Background] Theodore WH, Spencer SS, Wiebe S, Langfitt JT, Ali A, Shafer PO, Berg AT, Vickrey BG. Epilepsy in North America: a report prepared under the auspices of the global campaign against epilepsy, the International Bureau for Epilepsy, the International League Against Epilepsy, and the World Health Organization. Epilepsia. 2006 Oct;47(10):1700-22. doi: 10.1111/j.1528-1167.2006.00633.x. PMID 17054693
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Pinti P, Siddiqui MF, Levy AD, Jones EJH, Tachtsidis I. An analysis framework for the integration of broadband NIRS and EEG to assess neurovascular and neurometabolic coupling. Sci Rep. 2021 Feb 17;11(1):3977. doi: 10.1038/s41598-021-83420-9. PMID 33597576
- [Background] Tremblay S, Rogasch NC, Premoli I, Blumberger DM, Casarotto S, Chen R, Di Lazzaro V, Farzan F, Ferrarelli F, Fitzgerald PB, Hui J, Ilmoniemi RJ, Kimiskidis VK, Kugiumtzis D, Lioumis P, Pascual-Leone A, Pellicciari MC, Rajji T, Thut G, Zomorrodi R, Ziemann U, Daskalakis ZJ. Clinical utility and prospective of TMS-EEG. Clin Neurophysiol. 2019 May;130(5):802-844. doi: 10.1016/j.clinph.2019.01.001. Epub 2019 Jan 19. PMID 30772238
- [Background] Grouiller F, Delattre BM, Pittau F, Heinzer S, Lazeyras F, Spinelli L, Iannotti GR, Seeck M, Ratib O, Vargas MI, Garibotto V, Vulliemoz S. All-in-one interictal presurgical imaging in patients with epilepsy: single-session EEG/PET/(f)MRI. Eur J Nucl Med Mol Imaging. 2015 Jun;42(7):1133-43. doi: 10.1007/s00259-015-3045-2. Epub 2015 Apr 17. PMID 25893383